CLINICAL TRIAL: NCT04544969
Title: Detecting Chemosensitivity and Predicting Treatmemt Efficacy With Circulating Tumour Cells From Peripheral Blood in Metastatic Nasopharyngeal Carcinoma Patients
Brief Title: Detecting Chemosensitivity and Predicting Treatmemt Efficacy With CTCs in mNPC
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, Prof., Sun Yat-sen University
Other Study IDs: B2019-128
Record Dates: First submitted 2020-08-03; First posted 2020-09-10 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Circulating Tumor Cell; Nasopharyngeal Carcinoma; Distant Metastases.Clinical; Effects of Chemotherapy
MeSH Terms: conditions — Neoplastic Cells, Circulating; Nasopharyngeal Carcinoma | interventions — Docetaxel; Cisplatin; Fluorouracil; Gemcitabine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chemotherapy: Patients treated with palliative chemotherapy
  Interventions: Drug: cisplatin-based chemotherapy

INTERVENTIONS:
Drug: cisplatin-based chemotherapy — GP: cisplatin 80 mg/m2 intravenous infusion on day1, gemcitabine 1000 mg/m2 intravenous infusion on day 1 and 8, both drugs are given every 3 weeks, recommended 6 cycles.
  TP: cisplatin 75 mg/m2 intravenous infusion in day1, docetaxel 75 mg/m2 intravenous infusion in day 1, both drugs are given every 3 weeks, recommended 6 cycles.
  PF: cisplatin 100 mg/m2 intravenous infusion in day1, fluorouracil 4000 mg/m2 intravenous infusion in day 1 to 5, both drugs are given every 3 weeks, recommended 6 cycles.
  TPF: cisplatin 60 mg/m2 intravenous infusion in day1, docetaxel 60 mg/m2 intravenous infusion in day 1, fluorouracil 3000 mg/m2 intravenous infusion in day 1 to 5, both drugs are given every 3 weeks, recommended 6 cycles.
  Choice of chemotherapy regimen is decided by patient's doctor in charge.
  Other Names: docetaxel and cisplatin; fluorouracil and cisplatin; docetaxel, fluorouracil and cisplatin; gemcitabine and cisplatin

SUMMARY:
The prospective observational clinical study will recruit 50 metastatic nasopharyngeal carcinoma (mNPC) patients, detecting patient's chemosensitivity with the circulating tumor cells (CTCs) from peripheral blood and prdicting patient's treatment efficacy with CTCs dynamic change.

ELIGIBILITY:
Inclusion Criteria:

* NPC patients with distant metastasis after 3 months of primary radiotherapy, and not suitable for local treatment
* At least having one measurable metastatic lesion
* All genders，range from 18～70 years old
* ECOG score 0 ~ 1
* Expected survival time ≥ 3 months
* White blood cell(WBC) count ≥ 3×109/L, neutrophile granulocyte(NE) count ≥ 1.5×109/L, hemoglobin(HGB) ≥ 90g/L, platelet(PLT) count ≥ 100×109/L
* Alanine aminotransferase (ALT) or aspartate aminotransferase(AST) < 2.5×upper limit of normal(ULN), bilirubin(BUN) or creatinine(CRE) < 1.5×ULN, alanine aminotransferase (CCR) ≥ 60ml/min
* Inform consent form

Exclusion Criteria:

* Have or are suffering from other malignant tumors;
* Participating in other clinical trials;
* Drug or alcohol addition;
* Do not have full capacity for civil acts;
* Mental disorder;
* Pregnancy or lactation;
* Severe complication, eg, uncontrolled hypertension.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NPC patients with distant metastasis after 3 months of primary radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The coincidence rate between drug sensitivity test in CTCs and objective response rate | 6 months
  Comparison the coincidence rate between drug sensitivity test in CTCs and objective response rate of corresponding chemotherapy regime

SECONDARY OUTCOMES:
The changes of CTCs countings | Change from pre-chemotherapy to 22-28(±7) days after last course of chemotherapy
Objective response rate | study period of 19 Months
  To be determined by measurement of target lesions according to RECIST criteria
Progression free survival | baseline
  Defined as the time in months from first course of treatment until PD is observed or death occurs due to any cause.
Cutoff value of CTC counts | Objective response at 6 months
  to identify patients with early relapse (<6 months) after liver resection as determined by the AUC under the ROC curve
Predictive value of the changes of CTCs countings | Change from pre-chemotherapy to 22-28(±7) days after last course of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn